CLINICAL TRIAL: NCT01323751
Title: A Phase 1/2, Open-Label, Multicenter Study of ACY-1215 Administered Orally as Monotherapy and in Combination With Bortezomib and Dexamethasone for the Treatment of Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Study of ACY-1215 Alone and in Combination With Bortezomib and Dexamethasone in Multiple Myeloma
Acronym: ACY-1215
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACY-100
Record Dates: First submitted 2011-02-25; First posted 2011-03-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ricolinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treat Regimen (Experimental): ACY-1215 Bortezomib Dexamethasone
  Interventions: Drug: ACY-1215

INTERVENTIONS:
Drug: ACY-1215 — Liquid oral dose on Days 1-5 and 8-12 of 21-day treatment cycle
  Other Names: HDAC6 inhibitor

SUMMARY:
Phase 1(a & b): To evaluate the side effects and determine the best dose of oral ACY-1215 as monotherapy, and also in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma.

Phase 2a: To determine the objective response rate of oral ACY-1215 in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient has relapsed or relapsed/refractory MM with measurable disease parameters according to the International Myeloma Working Group (IMWG) Criteria

  * Refractory is defined as experiencing less than minimal response (MR) to or progressive disease (PD) within 60 days after completion of the most recent anti-MM regimen
  * Relapsed is defined as experiencing PD that requires therapy but which is not refractory following the achievement of stable disease (SD) or better to the most recent anti-MM regimen.
* Patient received at least 2 prior regimens for MM.
* Patient received prior treatment for MM with a proteasome inhibitor and an immunomodulatory drug, unless not a candidate for a proteasome inhibitor or an immunomodulatory drug.
* Patient either is not a candidate for autologous stem cell transplant (ASCT), has declined the option of ASCT, or has relapsed after prior ASCT.
* Patient is ≥18 years of age.
* Patient has a Karnofsky Performance Status score of ≥70
* Patient has adequate bone marrow reserve, as evidenced by:

  * Absolute neutrophil count (ANC) of ≥1.0x109/L.
  * Platelet count of ≥ 75x109/L in patients in whom <50% of bone marrow nucleated cells are plasma cells and ≥50x109/L in patients in whom more than 50% of bone marrow nucleated cells are plasma cells.
* Patient has adequate renal function (calculated creatinine clearance of ≥30 mL/min according to the Cockroft-Gault)
* Patient has adequate hepatic function (serum bilirubin values <2.0 mg/dL and ALT and/or AST values <3 × the upper limit of normal ULN).
* Patient has a corrected serum calcium ≤ULN.

Exclusion Criteria

* Patient has received any of the following therapies:

  * Radiotherapy or systemic therapy within 2 weeks of baseline
  * Prior peripheral autologous stem cell transplant within 12 wks of Baseline.
  * Prior allogeneic stem cell transplant.
  * Prior treatment with an HDAC inhibitor.
* Patient has an active systemic infection requiring treatment.
* Patient has a history of other malignancies unless has undergone definitive treatment more than 5 yrs prior to study and without evidence of recurrent malignant disease (excluding basal cell carcinoma of the skin; superficial carcinoma of the bladder; carcinoma of the prostate with a current prostate-specific antigen <0.1 ng/mL; or cervical intraepithelial neoplasia).
* Patient has known or suspected HIV, positive for hepatitis B or is known or suspected to have active hepatitis C infection.
* Patient has a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness including recent myocardial infarction (within 6 months)or stroke; hypertension requiring >2 medications for adequate control; diabetes mellitus with >2 episodes of ketoacidosis in the preceding 12 months; or chronic obstructive pulmonary disease (COPD) requiring >2 hospitalizations in the preceding 12 months.
* Patient has a QTcF value of >480 msec; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy; previous history of drug-induced QTc prolongation
* Patient has > Grade 2 painful neuropathy or peripheral neuropathy
* Patient has a history of allergic reaction attributable to bortezomib or other compounds containing boron or mannitol (Phase 1b and 2a only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12-03 (Actual)

PRIMARY OUTCOMES:
Phase 1 (a & b): To determine the maximum tolerated dose of ACY-1215 as monotherapy or in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma. | Upon completion of 21-day treatment cycle
Phase 2a: To determine the objective response rate to ACY-1215 in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma. | Assessed every other treatment cycle (cycles 2, 4 and 6)

SECONDARY OUTCOMES:
Characterize the safety of ACY-1215 alone or in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma | Up to 24 weeks
Determine the single- and multiple-dose PK of ACY-1215 alone and in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma | Upon completion of 21 day treatment cycle
Evaluate the pharmacodynamics of ACY-1215 alone or in combination with bortezomib and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma. | Up to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Lonial, MD, Principal Investigator — Winship Cancer Institute, Emory University
Locations (6):
- United States (6):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mt. Sinai Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin - Clinical Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes